CLINICAL TRIAL: NCT05921864
Title: Study of Biomarkers of Heat Tolerance and Recovery During Ultra-endurance Exercise
Acronym: PENTHERE
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PBMD05; 2023-A00730-45 (Other: IDRCB)
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Heat Stress; Heat
Keywords: ultra-endurance
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Passive heat exposure — Participants will be exposed to heat in a chamber.
Other: Active heat exposure — Participants will participate to a 6-hour run.

SUMMARY:
Military personnel are called upon to serve in hot, dry or humid climates, which places great demands on their ability to tolerate heat. Induced heat stress can impair performance and lead to pathologies. Faced with the challenges of global warming, this issue is becoming increasingly important in the practice of sport. While hyperthermia is known to impair endurance performance, the underlying thermophysiological responses and regulatory mechanisms during prolonged exercise remain poorly understood. The effects of hyperthermia on mental performance raise questions about the degradation of interoceptive capacities and the deleterious impact on behavioral regulation, an important component of thermal risk management in ultra-endurance exercise. What's more, despite the muscular and hydromineral consequences (rhabdomyolysis, renal failure, dehydration) of prolonged exercise, few data are available on recovery kinetics. A better understanding of the factors conditioning recovery quality could help limit the deleterious consequences of ultra-endurance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* BMI between 18 and 25 kg/m2
* Weight ≥ 51 kg
* Minimum training volume 6 days/7, aerobic
* Participation in a running competition ≥ 6hours
* Having given informed consent

Exclusion Criteria:

* Presence or history of medical pathology
* Presence of significant deviation from normal electrocardiogram values
* History of heat stroke
* Known intolerance to heat
* Inability to swallow a capsule or refusal of rectal probe
* Alcohol consumption exceeding the equivalent of 3 glasses of wine per week
* Consumption of narcotics
* Smoking > 0.5 pack of cigarettes per day
* On usual medication
* Pregnant or breast-feeding women
* Protected adult, under legal protection, guardianship or curatorship, or unable to give personal written consent

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be composed of healthy young athletes.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Degree of correlation between core temperature measured at the end of passive heat exposure and that measured at the end of active heat exposure | Through study completion (1 month)
  Core temperature will be measured in every participants at the end of passive heat exposure and at the end of active heat exposure. A correlation analysis will be performed on these measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided